CLINICAL TRIAL: NCT02000544
Title: Clinical Evaluation Study of a Novel Modular Extracorporeal Circulation Circuit in Open Heart Surgery
Brief Title: Clinical Evaluation of a Modular Extracorporeal Circulation Circuit
Acronym: MiECC MODULAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AHEPA University Hospital (Other)
Responsible Party: Principal Investigator, Kyriakos Anastasiadis, Professor Kyriakos Anastasiadis, AHEPA University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MiECC MODULAR
Record Dates: First submitted 2013-10-06; First posted 2013-12-04 (Estimated); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Coronary Artery Disease; Aortic Valve Disease; Mitral Valve Disease; Aortic Aneurysm
Keywords: Extracorporeal Circulation; Cardiopulmonary Bypass; Cardiac surgery
MeSH Terms: conditions — Coronary Artery Disease; Aortic Valve Disease; Aortic Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Modular Cardiopulmonary Bypass Circuit (Other): Patients undergoing open heart surgery with a modular hybrid extracorporeal circulation circuit.
  Interventions: Device: Modular Cardiopulmonary Bypass Circuit

INTERVENTIONS:
Device: Modular Cardiopulmonary Bypass Circuit — Open heart surgery with a novel hybrid modular extracorporeal circulation circuit which is a closed cardiopulmonary bypass circuit with enhanced safety as it can be instantly converted to an open circuit.

SUMMARY:
The purpose of this clinical research study is the design of a novel modular hybrid system extracorporeal circulation circuit for open heart procedures that could easily be converted from a closed to a semi-closed circuit according to the indication. This could expand the potential of minimal extracorporeal circulation and could ultimately become the new standard circuit in performing every type of cardiac surgery.

DETAILED DESCRIPTION:
Development of cardiopulmonary bypass circuit (heart-lung machine) is considered as a landmark breakthrough in cardiac surgery, greatly promoting treatment of cardiovascular diseases. Since 1953, when the first operation under cardiopulmonary bypass was performed and for almost 6 decades, little progress has been made in the direction of improving cardiopulmonary bypass technology. However, evolution is feasible. The proposed research project challenges the traditional belief that conventional cardiopulmonary bypass should be considered as "state of the art" technology by deducting solid evidence towards extended use of the novel minimal extracorporeal circulation circuit, which is related to an improved outcome through multiple studies. Research methodology is based on analyzing laboratory and clinical data obtained through implementing the standard and the novel technology. In order to provide solid evidence on the comparative effectiveness of both therapies, it combines analysis of clinical and laboratory data with data related to cost and quality of life. Thus, it assesses novel technology from a global perspective and the evidence obtained would be considered robust.

The ultimate purpose of the research proposal is the design of a modular hybrid system, that could easily convert from form a closed to a semi-closed circuit according to the indication, that could expand the potential of minimal extracorporeal circulation and could ultimately become the new standard circuit in performing every type of cardiac surgery. The term modular refers to an additionally mounted, clamped-off venous reservoir which allows to run the system as an open circuit in case of anticipated volume loss (ie bleeding, complex procedures, long bypass run). This measure follows the proverb 'always expect the unexpected' and offers the clinical practitioner an additional safety margin in case of unexpected intraoperative events. Unique design of this circuit would offer the opportunity of reducing cost, while at the same time improving clinical outcome. Preliminary design of this circuit, performed in our institution, is presented schematically in the appendix. After completion of the study protocol the designed circuit will be patented.

Our institution has already performed extensive research and has gained international reputation as a training centre on minimal extracorporeal circulation. Design of such a circuit could promote further research funded by the medical industry. Considering the number of cardiac surgical procedures performed every day worldwide, this evolution is greatly ambitious and could be characterized as a major breakthrough in the field of cardiac surgery opening up new horizons in the field of cardiovascular research. It would also exert a positive effect on global healthcare affecting lives of millions of people suffering from cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Any heart disease that requires open heart surgery under extracorporeal circulation

Exclusion Criteria:

* Beating heart surgery
* Age more than 80 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2013-10; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Rate of conversion to an open circuit | Intraoperartive
  Conversion rate from closed type-III MiECC to an open circuit

CONTACTS AND LOCATIONS:
Overall Officials: Kyriakos Anastasiadis, MD, DSc, FETCS, Study Director — AHEPA University Hospital
Locations (1):
- AHEPA University Hospital, Thessaloniki, Greece

REFERENCES:
- [Background] Anastasiadis K, Fragoulakis V, Antonitsis P, Maniadakis N. Coronary artery bypass grafting with minimal versus conventional extracorporeal circulation; an economic analysis. Int J Cardiol. 2013 Oct 15;168(6):5336-43. doi: 10.1016/j.ijcard.2013.08.006. Epub 2013 Aug 15. PMID 23992927
- [Background] Anastasiadis K, Asteriou C, Antonitsis P, Argiriadou H, Grosomanidis V, Kyparissa M, Deliopoulos A, Konstantinou D, Tossios P. Enhanced recovery after elective coronary revascularization surgery with minimal versus conventional extracorporeal circulation: a prospective randomized study. J Cardiothorac Vasc Anesth. 2013 Oct;27(5):859-64. doi: 10.1053/j.jvca.2013.01.010. Epub 2013 Jun 18. PMID 23791499
- [Background] Asteriou C, Antonitsis P, Argiriadou H, Deliopoulos A, Konstantinou D, Foroulis C, Papakonstantinou C, Anastasiadis K. Minimal extracorporeal circulation reduces the incidence of postoperative major adverse events after elective coronary artery bypass grafting in high-risk patients. A single-institutional prospective randomized study. Perfusion. 2013 Jul;28(4):350-6. doi: 10.1177/0267659113479135. Epub 2013 Mar 21. PMID 23520169
- [Background] Anastasiadis K, Antonitsis P, Haidich AB, Argiriadou H, Deliopoulos A, Papakonstantinou C. Use of minimal extracorporeal circulation improves outcome after heart surgery; a systematic review and meta-analysis of randomized controlled trials. Int J Cardiol. 2013 Apr 5;164(2):158-69. doi: 10.1016/j.ijcard.2012.01.020. Epub 2012 Feb 8. PMID 22325958
- [Background] Anastasiadis K, Antonitsis P, Argiriadou H, Khayat A, Papakonstantinou C, Westaby S. Use of minimal extracorporeal circulation circuit for left ventricular assist device implantation. ASAIO J. 2011 Nov-Dec;57(6):547-9. doi: 10.1097/MAT.0b013e318232d5d5. PMID 21970982
- [Background] Anastasiadis K, Chalvatzoulis O, Antonitsis P, Deliopoulos A, Argiriadou H, Karapanagiotidis G, Kambouroglou D, Papakonstantinou C. Use of minimized extracorporeal circulation system in noncoronary and valve cardiac surgical procedures-a case series. Artif Organs. 2011 Oct;35(10):960-3. doi: 10.1111/j.1525-1594.2010.01183.x. Epub 2011 Apr 19. PMID 21501191
- [Background] Anastasiadis K, Argiriadou H, Kosmidis MH, Megari K, Antonitsis P, Thomaidou E, Aretouli E, Papakonstantinou C. Neurocognitive outcome after coronary artery bypass surgery using minimal versus conventional extracorporeal circulation: a randomised controlled pilot study. Heart. 2011 Jul;97(13):1082-8. doi: 10.1136/hrt.2010.218610. Epub 2011 Feb 28. PMID 21357641
- [Background] Anastasiadis K, Westaby S, Antonitsis P, Argiriadou H, Karapanagiotidis G, Pigott D, Papakonstantinou C. Minimal extracorporeal circulation circuit standby for "off-pump" left ventricular assist device implantation. Artif Organs. 2010 Dec;34(12):1156-8. doi: 10.1111/j.1525-1594.2009.00983.x. PMID 20545669
- [Background] Anastasiadis K, Asteriou C, Deliopoulos A, Argiriadou H, Karapanagiotidis G, Antonitsis P, Grosomanidis V, Misias G, Papakonstantinou C. Haematological effects of minimized compared to conventional extracorporeal circulation after coronary revascularization procedures. Perfusion. 2010 Jul;25(4):197-203. doi: 10.1177/0267659110373840. Epub 2010 Jun 1. PMID 20515982